CLINICAL TRIAL: NCT02968160
Title: A Clinical Trial of YMC017 in Hypertensive and Hypercholesterolemic Patients With Metabolic Syndrome
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to poor enrollment rate
Sponsor: Yuhan Corporation (Industry)
Collaborators: Linical Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMC017
Record Dates: First submitted 2016-11-10; First posted 2016-11-18 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2017-05

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Telmisartan; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telmisartan+Rosuvastatin (Experimental): Duowell ® tablet (Telmisartan 40mg + Rosuvastatin 20mg) 1 tablet, once daily, Oral administration/ 8 weeks
  * But, the increased Duowell ® tablet (Telmisartan 80mg + Rosuvastatin 20mg) will get administrated orally one tablet once daily to the subjects who have mean systolic blood pressure more than 140mmHg based on arm, which was determined before, at 4week visit.
  Interventions: Drug: Telmisartan 40mg + Rosuvastatin 20mg; Drug: Telmisartan 80mg + Rosuvastatin 20mg
- Telmisartan/Rosuvastatin (Active Comparator): Telmisartan 40mg + Rosuvastatin 20mg 2 tablets, once daily, Oral administration/ 8 weeks
  * But, the increased Telmisartan 80mg + Rosuvastatin 20mg will get administrated orally 2 tablets once daily to the subjects who have mean systolic blood pressure more than 140mmHg based on arm, which was determined before, at 4week visit.
  Interventions: Drug: Telmisartan 40mg, 80 mg; Drug: Rosuvastatin 20mg

INTERVENTIONS:
Drug: Telmisartan 40mg + Rosuvastatin 20mg
  Other Names: Duowell ® tablet
  Arms: Telmisartan+Rosuvastatin
Drug: Telmisartan 80mg + Rosuvastatin 20mg
  Other Names: Duowell ® tablet
  Arms: Telmisartan+Rosuvastatin
Drug: Telmisartan 40mg, 80 mg
  Other Names: Micardis tablet
  Arms: Telmisartan/Rosuvastatin
Drug: Rosuvastatin 20mg
  Other Names: Monorova tablet
  Arms: Telmisartan/Rosuvastatin

SUMMARY:
This is a Randomized, open-label, 2 groups, parallel design.

DETAILED DESCRIPTION:
This study objective is to compare the safety and efficacy between fixed dose combination (Duowell® tab) and free pill combination therapy of Telmisartan and Rosuvastatin in hypertensive and hypercholesterolemic patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 19 and 79 years old at screening visit
* Subjects who have being used anti-hypertension drugs and Lipid lowering agents over 4weeks before randomization.
* Subjects who have been diagnosed with metabolic syndrome according to following criteria Definition of patients with metabolic syndrome: Patients satisfy two of the following criteria at least

  * Abdominal obesity: Waist measurement > 90 cm(male), > 80 cm(female)
  * Triglyceride(TG) ≥ 150 mg/dL(
  * High-Density Lipoprotein Cholesterol(HDL-C) < 40 mg/dL(male), < 50 mg/dL (female)
  * Fasting Plasma Glucose(FPG) ≥ 100 mg/dL or Subject who has being used oral hypoglycemic agents
* Childbearing potential women have certainly negative of the pregnancy test at screening visit (visit 1), and agree to implement the effective contraception during the study period(including the medically non-pregnant state)
* Subjects who have signed after fully understanding the purpose, content, characteristics and risk of the investigational product and get explained enough.

Exclusion Criteria:

* Subjects who taking anti-hypertension drugs more than three agent
* Subjects who have mean Sitting Systolic Blood Pressure(siSBP) > 160 mmHg (excluded if appliable, one of the arms)
* Subjects who have blood pressure ≥ 140/90 mmHg with taking 2 or more anti-hypertension drugs (except if any of the arms)
* Subjects that Low Density Lipoprotein-Cholesterol(LDL-C) isn't properly controlled according to National Cholesterol Education Program Adults Treatment Panel (NCEP ATP) III criteria
* Subjects who have triglyceride (TG) ≥ 400mg/dL
* Subjects who have a difference more than 20mmHg at the mean Sitting Diastolic Blood Pressure(siSBP) measured three times in both arms.
* Other exclusions applied

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-10; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects that the mean Sitting Diastolic Blood Pressure(siSBP) and Low Density Lipoprotein-Cholesterol(LDL-C) level reach the treatment goals after 8 weeks from investigational product administration. | week 8

SECONDARY OUTCOMES:
Change of Low Density Lipoprotein-Cholesterol(LDL-C) from baseline to 4 and 8 weeks | From baseline to 4 and 8 weeks
Change of Sitting Systolic Blood Pressure(siSBP) and Sitting Diastolic Blood Pressure(siDBP) from baseline to 4 and 8 weeks | From baseline to 4 and 8 weeks
The proportion of subjects that the mean sitting blood pressure(siBP) level reaches the treatment goals to 4 and 8 weeks | 4 and 8 weeks
The proportion of subjects that the Low Density Lipoprotein-Cholesterol(LDL-C) level reaches treatment goals in accordance with guideline of National Cholesterol Education Program-Adult Treatment Panel(NCEP ATP) III to 4 and 8 weeks | 4 and 8 weeks
Change of below indicators from baseline to 4 and 8 weeks | baseline to 4 and 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguk University Medical Center, Ilsan, South Korea

IPD SHARING:
Plan to Share IPD: No